CLINICAL TRIAL: NCT03062306
Title: Can Sufficient Cerebral Oxygenation be Provided in a Synchronized Manner With Chest Compression During Cardiopulmonary Resuscitation?
Brief Title: Chest Compression and Cerebral Oxygenation During Cardiopulmonary Resuscitation
Acronym: CPR
Status: Completed | Type: Observational
Sponsor: Nevsehir Public Hospital (Other Government)
Responsible Party: Principal Investigator, Mehmet Akif Yazar, Critical Care Physician, Nevsehir Public Hospital
Other Study IDs: 2016/351; Erciyes University (Other: Clinical Research Ethics Committee)
Record Dates: First submitted 2017-02-16; First posted 2017-02-23 (Actual); Last update posted 2019-02-22 (Actual); Status verified 2019-02

CONDITIONS: Providing Sufficient Cerebral Oxygenation During CPR
Keywords: Cerebral Oxygenation; Cardiopulmonary Resuscitation; Chest Compression

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In recent years, monitorizations during Cardiopulmonary Resuscitation (CPR) are inadequate to show the sufficiency of cerebral oxygenation. During CPR, insufficient chest compressions have critical importance for neurological results and life quality after the return of spontaneous circulation (ROSC).

DETAILED DESCRIPTION:
The Near-Infrared Spectroscopy (NIRS), which is used in measuring the cerebral tissue oxygenation is one of the latest technologies that allow the measurement of brain oxygen saturation. With this study, the issue of whether sufficient cerebral oxygenation is provided during CPR applied to patients that have Cardiac Arrest (CA) will be investigated, and the effect of CPR on the patient prognosis after ROSC will be examined. In this study, the aim is to investigate whether sufficient oxygenation is provided in synchronization with chest compressions during CPR; and to test the regional brain tissue saturation with rSO2 measurement, and the prognosis with Full Outline of UnResponsiveness (FOUR) Score in patients with ROSC.

ELIGIBILITY:
Inclusion Criteria:

1. All patients undergoing cardiac arrest in intensive care unit

Exclusion Criteria:

1. Head injury and intracranial bleeding
2. Cerebral ischemic vascular event
3. Pulmonary diseases that may affect blood-oxygen levels
4. Below the age of 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients undergoing cardiac arrest in intensive care unit
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2017-05-31 (Actual); Primary Completion 2017-08-31 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
The levels of regional brain tissue oxygen saturation (rSO2) providing with chest compressions during Cardiopulmonary Resuscitation (CPR) | About six month
  The data will be obtained by using the Near Infrared Spectroscopy (NIRS) Device and will be recorded rSO2 measurement during the resuscitation of the Cardiac Arrest (CA) patients

SECONDARY OUTCOMES:
Change from baseline in consciousness on Full Outline of UnResponsiveness (FOUR) Score at one week | For a week after ROSC
  The patient's consciousness will be evaluated by FOUR score in patients with ROSC

CONTACTS AND LOCATIONS:
Locations (1):
- Mehmet Akif YAZAR, Nevşehir, Turkey (Türkiye)

REFERENCES:
- [Background] Parnia S, Nasir A, Shah C, Patel R, Mani A, Richman P. A feasibility study evaluating the role of cerebral oximetry in predicting return of spontaneous circulation in cardiac arrest. Resuscitation. 2012 Aug;83(8):982-5. doi: 10.1016/j.resuscitation.2012.01.039. Epub 2012 Feb 6. PMID 22322284
- [Background] Kamarainen A, Sainio M, Olkkola KT, Huhtala H, Tenhunen J, Hoppu S. Quality controlled manual chest compressions and cerebral oxygenation during in-hospital cardiac arrest. Resuscitation. 2012 Jan;83(1):138-42. doi: 10.1016/j.resuscitation.2011.09.011. Epub 2011 Sep 28. PMID 21958930